CLINICAL TRIAL: NCT01068236
Title: Primary Care Treatment for Overweight Adolescent Females
Brief Title: Primary Care Treatment for Overweight Adolescent Females (SHINE)
Acronym: SHINE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Victor J. Stevens, PhD /Senior Investigator, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R01HD050931-04 (NIH); NCT00451685 (obsolete NCT alias)
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-03

CONDITIONS: Obesity
Keywords: Teen girls; weightloss; healthy lifestyle; yoga; Weight loss and healthy lifestyle
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy lifestyle intervention (Experimental): lifestyle/weight-loss intervention for overweight (95th - 99th percentile) female adolescents (13-15 years of age at study entry) to a usual-care control condition. The intervention will be 20-sessions and combines group visits, individual telephone coaching calls, and tailored pediatric primary care providers (PCP) visits.
  Interventions: Behavioral: Healthy lifestyle managment
- Usual care (No Intervention): In the usual care control condition adolescents and their family will receive individualized feedback from the assessments as well as handouts outlining healthy means of maintaining / reducing weight for adolescents through improving nutrition and physical activity. In addition, these participants will be encouraged to seek any appropriate health care/education services available through Kaiser Permanente or in the community.

INTERVENTIONS:
Behavioral: Healthy lifestyle managment — Exercise, yoga, food diaries, provider consultation
  Arms: Healthy lifestyle intervention

SUMMARY:
This project will examine the effectiveness of a primary care based intervention to help overweight teen girls adopt healthy lifestyle practices. Participants are adolescent females at select Kaiser Permanente Northwest primary care clinics with a body mass index above the 90th percentile. Teens will be randomly assigned to (1) a behavioral weight control program (enriched intervention), (or 2) usual-care (control). Primary care providers of teens in the intervention condition are given customized plans describing the teen's eating and physical activity habits and instructions on how to best work with these teens and their families. The behavioral weight control program is specifically tailored for teen girls and includes separate group meetings for teens and parents, follow-up telephone contacts with their group leader, and coordinated feedback from the teen's primary care provider.

DETAILED DESCRIPTION:
Obesity is currently a major US public health problem, given its prevalence and adverse health consequences. In the past two decades, the percentage of overweight adolescents has almost tripled from 5 to 14%. Clinic-based weight control treatments for youth have demonstrated some success, but most have been designed for pre-adolescent children and their families. Even though considerable research explores adult-weight control and a growing body of research examines childhood obesity, treatments for adolescents have not been adequately studied. Also, almost all empirically tested interventions for youth have been based in academic research clinics rather than in primary care medical settings, where weight problems are most often identified and may be most efficiently treated. Placing adolescent weight-related interventions in primary medical care settings could make them both more easily disseminated and more cost-effective. Finally, treating obesity in a primary care (non-school) setting may be particularly effective/appropriate for teen girls for two reasons. First, overweight girls are at higher risk than normal-weight peers for engaging in unhealthy weight-control behaviors. Second, researchers speculate that teen girls' self-consciousness in mixed-gender physical education (PE) classes may contribute to their lower enrollment rates enrollment in PE classes and overall decline in physical activity in recent years. If so, targeting physical activity in a primary-care-based program may be more successful than in school-based programs.

We propose to examine the clinical effectiveness and incremental cost-effectiveness of a primary care-based multi-component lifestyle intervention for overweight adolescent females and their families. This multi-component intervention will be tailored for gender and developmental stage, and will include a behaviorally-based intervention for teens and parents as well as coordinated feedback and counseling from the adolescent's pediatric primary care provider (PCP). We will compare the primary care-based intervention to a usual-care control condition in which adolescents and their family receive information about weight loss and guidelines for achieving and maintaining a healthy lifestyle along with the encouragement to utilize any appropriate health care services.

The principal aim of the study is to determine the clinical effectiveness of a primary care-based, multi-component lifestyle intervention for overweight (≥ 90th percentile) adolescent females and their families. H1: We hypothesize that the treatment group will have a greater decrease in BMI z-score from baseline to 12 months than the control youth.

In addition, we include the following secondary aims that are exploratory and intended to be hypothesis-generating rather than hypothesis-testing activities:

Determine if dietary intake (total energy intake, % calories from fat, etc.) and/or physical activity mediate the effect of the intervention on BMI z score. H2: Change in dietary intake and physical activity from baseline to 6 months will mediate the relationship between the intervention and change in BMI z score from baseline to 12 months.

Determine the impact of the experimental intervention for overweight adolescents and their families on the secondary outcomes including other physiological parameters (triglycerides, cholesterol, fasting insulin), quality of life, and psychosocial functioning; participant safety (depression and disordered eating behaviors); and feasibility/acceptability of the intervention (e.g., participant and provider satisfaction) in preparation for future Phase III trials.

Determine the incremental cost-effectiveness of the intervention relative to usual care from the societal perspective. We will examine the direct cost of delivering the intervention and this treatment's impact on subsequent use and cost of health services. We also will include indirect costs to participants and their families due to their participation in the intervention and use of other health care services (e.g., time spent in travel, usual care visits, out-of session activities).

ELIGIBILITY:
Inclusion Criteria:

* Females,
* Ages 13- 15 at study recruitment,
* BMI in overweight range (95th percentile - 99th percentile,
* One or both parent(s) willing to participate.

Exclusion Criteria:

* BMI > 99th percentile,
* Significant cognitive impairment,
* Current pregnancy,
* Congenital heart disease that limits activity,
* Serious asthma requiring oral prednisone,
* Taking medications that increase appetite.

Ages: 13 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 215 (Actual)
Dates: Start 2005-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
BMI z-score | 2 years

SECONDARY OUTCOMES:
Blood pressure | One year
Fasting lipid profile | One year
Fasting glucose | One year

CONTACTS AND LOCATIONS:
Overall Officials: Victor J Stevens, PhD, Principal Investigator — Kaiser Permanente

REFERENCES:
- [Derived] DeBar LL, Stevens VJ, Perrin N, Wu P, Pearson J, Yarborough BJ, Dickerson J, Lynch F. A primary care-based, multicomponent lifestyle intervention for overweight adolescent females. Pediatrics. 2012 Mar;129(3):e611-20. doi: 10.1542/peds.2011-0863. Epub 2012 Feb 13. PMID 22331335